CLINICAL TRIAL: NCT01328275
Title: The Thai HIV Disease Progression: An Observational Database
Brief Title: Progress Adult Study
Status: Completed | Type: Observational
Sponsor: The HIV Netherlands Australia Thailand Research Collaboration (Other)
Collaborators: Bamrasnaradura Infectious Diseases Institute (Other Government); Sanpatong Hospital (Unknown)
Responsible Party: Sponsor
Other Study IDs: HIV-NAT 153
Record Dates: First submitted 2011-03-02; First posted 2011-04-04 (Estimated); Last update posted 2016-05-11 (Estimated); Status verified 2016-05

CONDITIONS: HIV; Depression
Keywords: HIV related adverse events; immunological failure; virological failure; quality of life; depression; genotypic resistance
MeSH Terms: conditions — Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: long-term follow-up of HIV-infected patients on ART
  Interventions: Drug: standard regimens according to the Thai Ministry of Public Health national guidelines

INTERVENTIONS:
Drug: standard regimens according to the Thai Ministry of Public Health national guidelines — Participants may receive any of the standard regimens. These regimens are recommended in the Thai Ministry of Public Health National guidelines for the treatment of HIV in children. Change of treatment will be according to the treating physicians.

SUMMARY:
The purpose of this study is to study the HIV disease progression in HIV-infected Thai Adult.

DETAILED DESCRIPTION:
This is a multicenter, observational prospective cohort study. All HIV-infected patients from Bamrasnaradura Institute, Sanpatong Hospital and HIV-NAT, Thai Red Cross AIDS Research Centre, are followed to assess HIV disease progression.

ELIGIBILITY:
Inclusion Criteria:

1. There is evidence that HIV infection true (blood positive results by ELISA (ELISA) has been confirmed or detected evidence co-infection. HIV in the body by PCR, HIV-RNA PCR).Currently on PI regimens
2. Signed consent form
3. Age> 18 years

Exclusion Criteria:

1. Patients who came for treatment in a department other than out patient, such as inpatient or emergency room.
2. Patients are not willing to receive treatment on a regular basis in all 3 hospitals as patients normally receive treatment at other hospitals on a regular basis. However, due to urgent events. Need to receive treatment in hospital and three of.
3. Patients who have been diagnosed by doctors as a Psychological disorder that can not store the data.
4. Patients who have been diagnosed by a medical condition that Alcoholism

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV-infected patients currently receiving ART at Bamrasnaradura Institute, Sanpatong Hospital or HIV-NAT, Thai Red Cross AIDS Research Centre, Bangkok.
Sampling Method: Probability Sample
Enrollment: 5600 (Actual)
Dates: Start 2007-12; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
HIV related adverse events | 1 year
  Time until patient has HIV related adverse events

SECONDARY OUTCOMES:
Immunological failure | 1 year
  time to immunological failure
virological failure | 1 year
  time to virological failure
the change of quality of life | 1 year
  time to change of quality of life
depression | 1 year
  time when patient develops depression
genotypic resistance | 1 year
  time to developing genotypic resistance

CONTACTS AND LOCATIONS:
Overall Officials: Wisit Prasithsirikul, MD, Principal Investigator — Bamrasnaradura infectious disease institute; Wirat Klinbuayam, MD, Principal Investigator — Sanpatong Hospital; Jintanat Ananworanich, MD, PhD, Principal Investigator — HIV-NAT, Thai Red Cross - AIDS Research Centre
Locations (3):
- Thailand (3):
  - Bamrasnaradura infectious disease institute, Nonthaburi, Changwat Nonthaburi
  - Sanpatong Hospital, Chiang Mai, Chiang Mai
  - HIV-NAT, Thai Red Cross AIDS Research Centre, Bangkok

REFERENCES:
- [Derived] Pongpirul W, Pongpirul K, Ananworanich J, Klinbuayaem V, Avihingsanon A, Prasithsirikul W. Chronic kidney disease incidence and survival of Thai HIV-infected patients. AIDS. 2018 Jan 28;32(3):393-398. doi: 10.1097/QAD.0000000000001698. PMID 29135575
- See also: HIV Netherlands Australia Thailand Research Collaboration (HIV-NAT) — http://www.hivnat.org